CLINICAL TRIAL: NCT00041288
Title: A Phase II Multicenter Randomized Study Of Two Non-Myeloablative Stem Cell Transplant Strategies For Low-Grade Lymphoma And Chronic Lymphocytic Leukemia (CLL)
Brief Title: Study Of Two Non-Myeloablative Stem Cell Transplant Strategies For Low-Grade Lymphoma And CLL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual and difficulty with multicenter logistics
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069462; UTSMC-0501228; AMGEN-UTSMC-0501228; IBMTR-SC-00-02.1; ROCHE-UTSMC-0501228; SPRI-UTSMC-0501228; NCI-V02-1706
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Leukemia; Lymphoma
Keywords: Waldenstrom macroglobulinemia; refractory chronic lymphocytic leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; Cyclosporine; fludarabine phosphate; Methotrexate; Mycophenolic Acid; Tacrolimus; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: methotrexate
Drug: mycophenolate mofetil
Drug: tacrolimus
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy. Sometimes the transplanted cells are rejected by the body's normal tissues. Cyclosporine, mycophenolate mofetil, methotrexate, and tacrolimus may prevent this from happening.

PURPOSE: Randomized phase II trial to compare the effectiveness of fludarabine plus total-body irradiation with that of combination chemotherapy followed by donor peripheral stem cell transplantation in treating patients who have relapsed non-Hodgkin's lymphoma or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the 1-year overall survival rate of patients with relapsed low-grade non-Hodgkin's lymphoma or chronic lymphocytic leukemia treated with fludarabine and total body irradiation vs cyclophosphamide and fludarabine followed by allogeneic peripheral blood stem cell transplantation and donor lymphocyte infusions.
* Compare the toxic effects of these regimens in these patients.
* Compare the incidence and severity of acute and chronic graft-versus-host disease in patients treated with these regimens.
* Compare the 1-year treatment-related mortality and infectious complications in patients treated with these regimens.
* Compare the efficacy of these treatment regimens, in terms of 1-year disease-free survival, of these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease, age (less than 55 vs over 55), and participating transplantation center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fludarabine IV on days -4 to -2. Patients undergo total body irradiation followed by allogeneic peripheral blood stem cell transplantation (PBSCT) on day 0. Patients receive graft-versus-host disease (GVHD) prophylaxis comprising oral cyclosporine twice daily on days -2 to 90 followed by a taper on days 90-150 and oral mycophenolate mofetil twice daily on days 0-28.
* Arm II: Patients receive fludarabine IV on days -6 to -2 and cyclophosphamide IV on days -3 to -2. Patients undergo PBSCT on day 0. Patients receive GVHD prophylaxis comprising methotrexate IV on days 1, 3, 6, and 11 and tacrolimus IV continuously and then orally on days -2 to 90 followed by a taper on days 90-150.

At approximately day 180, patients with persistent disease, evidence of T-cell chimerism, and no GVHD may receive up to 3 donor lymphocyte infusions administered every 1-2 months.

Quality of life is assessed at baseline, 1 month, every 3 months for 1 year, and then every 6 months for 1 year.

Patients are followed at 1 month, every 3 months for 1 year, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia or
* Diagnosis of non-Hodgkin's lymphoma
* Lymphoplasmacytic lymphoma
* Grade I follicular small cleaved cell lymphoma
* Grade II follicular mixed cell lymphoma
* Diffuse small cleaved cell lymphoma
* Small lymphocytic lymphoma
* Relapsed after at least 1 course of prior therapy
* Availability of a 6/6 human leukocyte antigen (HLA) A, B, and DR identical sibling donor
* Nonmyeloablative transplantation candidate
* No clinically significant effusions or ascites that would preclude administration of methotrexate

PATIENT CHARACTERISTICS:

-Age: 18 to 75

Performance status:

* Eastern Cooperative Oncology Group (ECOG) 0-2 OR Zubrod 0-2
* Life expectancy: At least 6 months
* Hematopoietic: Not specified
* Hepatic: Bilirubin no greater than 3 mg/dL
* Renal: Creatinine no greater than 2 mg/dL
* Cardiovascular: left ventricular ejection fraction (LVEF) at least 40% on multigated acquisition (MUGA) scan or echocardiogram
* Pulmonary: diffusing capacity of lung for carbon monoxide (DLCO) at least 50% of predicted

OTHER:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled bacterial, viral, fungal, or parasitic infection
* Human Immunodeficiency Virus (HIV)1 and Human Immunodeficiency Virus (HIV)2 negative
* No other active malignancy except basal cell skin cancer
* No recent history of drug or alcohol abuse
* No other primary disease or comorbid illness that would severely limit life expectancy

PRIOR CONCURRENT THERAPY

* Biologic therapy:See Disease Characteristics
* Biologic therapy:Prior autologous bone marrow transplantation allowed if disease has progressed after transplantation
* Biologic therapy:No entry on study as part of a tandem autologous transplantation followed by nonmyeloablative allograft protocol
* Chemotherapy: Not specified
* Endocrine therapy: Not specified
* Radiotherapy:Not specified
* Surgery: Not specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2001-10; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Collins, MD, Study Chair — Simmons Cancer Center
Locations (23):
- United States (19):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Delaware Clinical & Laboratory Physicians, Newark, Delaware
  - Florida Hospital Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Missouri Kansas City School of Medicine, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - James P. Wilmot Cancer Center, Rochester, New York
  - Oregon Cancer Institute, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Massey Cancer Center, Richmond, Virginia
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - University of Toronto, Toronto, Ontario
  - Hopital du Saint-Sacrament, Quebec, Québec, Quebec